CLINICAL TRIAL: NCT04140175
Title: A Multicenter, Observational Cohort Study of Women Receiving Standard of Care (SOC) for the Treatment of Pelvic Pain Attributable to Suspected or Confirmed Endometriosis
Brief Title: A Study of Women Receiving Standard of Care (SOC) for the Treatment of Pelvic Pain Due to Suspected or Confirmed Endometriosis and the Impact on the Disease or Symptom Progression.
Status: Terminated | Type: Observational
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-836
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Endometriosis; Chronic Pelvic Pain; Dysmenorrhea
Keywords: Endometriosis; Chronic Pelvic Pain; Dysmenorrhea
MeSH Terms: conditions — Endometriosis; Dysmenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women with suspected or confirmed endometriosis: Women with suspected or confirmed endometriosis undergoing standard of care treatments or interventions.

SUMMARY:
This study will describe historic, current, and evolving treatment pathways, treatments, and interventions in women with a suspected or confirmed diagnosis of endometriosis in order to better understand the impact of early intervention on the disease or its symptoms. Length of treatment is dependent on standard of care treatment provided and all study information will be collected during routine standard of care visits.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (between their first menstrual cycle and before onset of menopause).
* Women who have experienced chronic pelvic pain (CPP) and/or dysmenorrhea (DYS) for at least 6 months prior to enrollment without symptom improvement with non-steroidal anti-inflammatory drugs (NSAIDs) or hormone/medical treatment.
* Women with suspected or confirmed endometriosis (EM) at time of enrollment.
* Women with CPP and/or DYS impacting daily activities as determined by their treating physician.
* Able to read, understand and respond to patient questionnaires.
* Willing to sign a patient authorization and/or informed consent form (ICF) and agree to disclose personal health information.

NOTE: For pediatric patients, parental/guardian assent/ICF is also required.

Exclusion Criteria:

* Women with chronic pelvic pain (CPP) and/or dysmenorrhea(DYS) for reasons other than endometriosis (EM).
* Women who have had a hysterectomy and/or bilateral ovary removal (oophorectomy).
* Women who are pregnant or planning to become pregnant.
* Women currently using assisted reproductive technologies such as in vitro fertilization (IVF).
* Women with a history of, or current malignancy (with or without systemic chemotherapy) with the exception of basal cell carcinoma of the skin.
* Women who are currently participating in an interventional clinical trial.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll women of reproductive age (between first onset of menses and before onset of menopause) with a suspected or confirmed diagnosis of endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Percentage of participants using specific medications for the treatment of chronic pelvic pain (CPP) and/or dysmenorrhea (DYS) | From onset of CPP and/or DYS to up to 4 years following study enrollment.
  Data regarding medication use for CPP and/or DYS will be collected from participant medical records, health care provider questionnaires, and participant completed questionnaires.
Percentage of participants who underwent surgical interventions for the treatment of CPP and/or DYS | From onset of CPP and/or DYS to up to 4 years following study enrollment.
  Percentage of participants who underwent surgical interventions for the treatment of CPP and/or DYS at any point from onset of CPP and/or DYS and study completion.
Number of surgical interventions for the treatment of CPP and/or DYS | From onset of CPP and/or DYS to up to 4 years following study enrollment.
  Number of surgical interventions for the treatment of CPP and/or DYS.
Percentage of participants undergoing hysterectomy | From study enrollment (Week 0) to up to 4 years.
  Percentage of participants undergoing hysterectomy during study enrollment.
Percentage of participants undergoing infertility treatment | From study enrollment (Week 0) to up to 4 years.
  Percentage of participants undergoing infertility treatments during study enrollment.
Percentage of participants undergoing surgery | From study enrollment (Week 0) to up to 4 years.
  Percentage of participants undergoing surgery as treatment for CPP and/or DYS.
Percentage of participants with complications associated with surgery | From study enrollment (Week 0) to up to 4 years.
  Percentage of participants with complications associated with surgery.
Percentage of participants receiving specific treatment sequences for the treatment of CPP and/or DYS | From onset of CPP and/or DYS to up to 4 years following study enrollment.
  Treatment sequences will be identified from the data. Treatment switching, add-on treatment, and discontinuations (including reasons) will be collected wherever possible.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (117):
- United States (117):
  - University of Alabama at Birmingham - Women's and Infant's Center /ID# 216236, Birmingham, Alabama
  - Atlanta VAMC /ID# 215763, Decatur, Alabama
  - Brown, Pearson, Guepet Gynecology /ID# 215500, Fairhope, Alabama
  - Women's Health Alliance of Mobile /ID# 213719, Mobile, Alabama
  - Mobile, Ob-Gyn, P.C. /ID# 217761, Mobile, Alabama
  - Visions Clinical Research-Tucs /ID# 216352, Tucson, Arizona
  - Olympia Clinical Trials /ID# 216238, Los Angeles, California
  - Camran Nezhat Institute /ID# 216083, Palo Alto, California
  - Infertility, Gynecology & Obst /ID# 213734, San Diego, California
  - West Coast Medical Research, I /ID# 217638, San Diego, California
  - Women's Care Clinic - Denver Health Main Campus /ID# 217975, Denver, Colorado
  - Advanced Women's Health Institute /ID# 217342, Greenwood Village, Colorado
  - Yale University /ID# 217978, New Haven, Connecticut
  - Stamford Hospital /ID# 216975, Stamford, Connecticut
  - Christiana Care Health Service /ID# 218097, Newark, Delaware
  - Reproductive Assoc of Delaware /ID# 216082, Newark, Delaware
  - Women's Medical Research Group /ID# 216230, Clearwater, Florida
  - GYN Research Institute - Kissimmee /ID# 217979, Kissimmee, Florida
  - Altus Research, Inc /ID# 213740, Lake Worth, Florida
  - South Florida Wellness & Clinic /ID# 217637, Margate, Florida
  - University of Miami /ID# 217952, Miami, Florida
  - Palmetto Professional Research /ID# 218051, Miami, Florida
  - A Premier Clinical Research of Florida, LLC /ID# 217949, Orange City, Florida
  - Physician Care Clin. Res., LLC /ID# 216570, Sarasota, Florida
  - GCP Clinical Research, LLC /ID# 218861, Tampa, Florida
  - University of South Florida /ID# 217606, Tampa, Florida
  - Stedman Clinical Trials /ID# 217595, Tampa, Florida
  - Journey Medical Research Insti /ID# 216077, Alpharetta, Georgia
  - Agile Clinical Research Trials /ID# 217762, Atlanta, Georgia
  - Academia Women's Health /ID# 218075, Atlanta, Georgia
  - Emory Saint Joseph's Hospital /ID# 213746, Atlanta, Georgia
  - Atlanta Women's Research Inst /ID# 216571, Atlanta, Georgia
  - Medisense Inc /ID# 218342, Atlanta, Georgia
  - Augusta OB/GYN Specialists LLC /ID# 218076, Augusta, Georgia
  - Paramount Research Solutions - College Park /ID# 217959, College Park, Georgia
  - WellStar Kennestone Women's Health Clinic /ID# 216983, Marietta, Georgia
  - Leavitt Womens Healthcare /ID# 221355, Idaho Falls, Idaho
  - Womens Healthcare Assoc, DBA /ID# 217839, Idaho Falls, Idaho
  - Advanced Clinical Research /ID# 218346, Meridian, Idaho
  - Women's Health Practice, LLC /ID# 216964, Champaign, Illinois
  - Northwestern Medicine Fertility and Reproductive Medicine /ID# 217662, Chicago, Illinois
  - Affinity Clinical Research /ID# 218203, Oak Brook, Illinois
  - The Advanced Gynecologic Surgery Institute - Park Ridge /ID# 217635, Park Ridge, Illinois
  - Women's Health Advantage /ID# 217951, Fort Wayne, Indiana
  - UnityPoint Clinic OB/GYN - Waterloo /ID# 216087, Waterloo, Iowa
  - Univ Kansas Med Ctr /ID# 216086, Kansas City, Kansas
  - Womens & Family Care, LLC dba /ID# 216569, Shawnee Mission, Kansas
  - Cypress Medical Research Ctr /ID# 218054, Wichita, Kansas
  - Norton Children's Gynecology /ID# 215671, Louisville, Kentucky
  - Horizon Research Group /ID# 217337, Eunice, Louisiana
  - Ochsner Baptist Medical Centre /ID# 215762, New Orleans, Louisiana
  - LSUHSC - Shreveport /ID# 216229, Shreveport, Louisiana
  - Omni Fertility and Laser Insti /ID# 217764, Shreveport, Louisiana
  - MaineGeneral Obstetrics & Gynecology /ID# 217634, Augusta, Maine
  - University of Maryland Med Ctr /ID# 216080, Baltimore, Maryland
  - Johns Hopkins University /ID# 217958, Baltimore, Maryland
  - Womens Health Center /ID# 216235, Glen Burnie, Maryland
  - Capital Women's Care - Hagerstown /ID# 217984, Hagerstown, Maryland
  - Boston Medical Center /ID# 218344, Boston, Massachusetts
  - Hanjani PC /ID# 217953, Brockton, Massachusetts
  - Boston Urogynecology Associates /ID# 216232, Cambridge, Massachusetts
  - NECCR Fall River LLC /ID# 216079, Fall River, Massachusetts
  - UMass Memorial Health Care /ID# 217608, Worcester, Massachusetts
  - Great Lakes Research, Inc. /ID# 215764, Bay City, Michigan
  - Central Michigan University Health /ID# 216237, Saginaw, Michigan
  - Saginaw Valley Med Res Group /ID# 217763, Saginaw, Michigan
  - University of Mississippi Medi /ID# 217636, Jackson, Mississippi
  - Saint Louis University School of Medicine /ID# 217633, St Louis, Missouri
  - CHI Health /ID# 216074, Omaha, Nebraska
  - R. Garn Mabey Jr, MD Chartered /ID# 218065, Las Vegas, Nevada
  - Cooper University Hospital/Sheridan Pavilion /ID# 218066, Marlton, New Jersey
  - Jersey Shore University Medical Center /ID# 216488, Neptune City, New Jersey
  - Rutgers Robert Wood Johnson /ID# 216972, New Brunswick, New Jersey
  - Circuit Clinical - Buffalo /ID# 217656, Buffalo, New York
  - Widewaters Gynecology /ID# 217661, East Syracuse, New York
  - Manhattan Medical Research /ID# 217950, New York, New York
  - Mount Sinai Medical Center - NY /ID# 216208, New York, New York
  - Suffolk Obstetrics and Gyneco /ID# 213781, Port Jefferson, New York
  - Richmond OB/GYN Associates PC /ID# 217642, Staten Island, New York
  - Island Reproductive Services - Staten Island /ID# 218202, Staten Island, New York
  - SUNY Upstate Medical University - Downtown /ID# 217596, Syracuse, New York
  - MAHEC OB/GYN Specialists /ID# 216973, Asheville, North Carolina
  - Carolina Women's Research and Wellness Center /ID# 216962, Durham, North Carolina
  - UNC Hospitals - Hillsborough /ID# 218343, Hillsborough, North Carolina
  - Eastern Carolina Women's Centr /ID# 217335, New Bern, North Carolina
  - M3 Wake Research Inc. /ID# 217167, Raleigh, North Carolina
  - Univ of Cincinnati Physicians /ID# 217643, Cincinnati, Ohio
  - University Hospitals Cleveland /ID# 216075, Cleveland, Ohio
  - MetroHealth Medical Center /ID# 217169, Cleveland, Ohio
  - Aventiv Research, Inc. /ID# 221293, Columbus, Ohio
  - Complete Healthcare for Women /ID# 216961, Columbus, Ohio
  - Wright State Univ, School Med /ID# 216084, Dayton, Ohio
  - Abington Reproductive Medicine /ID# 216575, Abington, Pennsylvania
  - Penn State University and Milton S. Hershey Medical Center /ID# 213787, Hershey, Pennsylvania
  - Vista Clinical Research /ID# 213789, Columbia, South Carolina
  - University Medical Group /ID# 217954, Greenville, South Carolina
  - Venus Gynecology, LLC /ID# 213790, Myrtle Beach, South Carolina
  - Palmetto Clinical Research /ID# 216076, Summerville, South Carolina
  - Women's Health Partners - Summerville /ID# 217339, Summerville, South Carolina
  - Chattanoogas Program in Womens /ID# 218052, Chattanooga, Tennessee
  - Chattanooga Medical Research /ID# 217594, Chattanooga, Tennessee
  - Paramount Research Solutions - Nashville /ID# 217341, Nashville, Tennessee
  - Urology Associates PC - Nashville /ID# 218139, Nashville, Tennessee
  - Methodist Dallas Medical Center /ID# 218350, Dallas, Texas
  - The Women's Centre /ID# 213794, Denton, Texas
  - Signature Gyn Services /ID# 216354, Fort Worth, Texas
  - Willowbend Health and Wellness - Frisco /ID# 217601, Frisco, Texas
  - Houston Methodist Hospital /ID# 216967, Houston, Texas
  - Univ Texas HSC San Antonio /ID# 218070, San Antonio, Texas
  - Physicians Research Options, L /ID# 213799, Draper, Utah
  - Granger Medical Clin-Riverton /ID# 218086, Riverton, Utah
  - Virginia Obstetrics & Gynecology /ID# 215797, Leesburg, Virginia
  - Virginia Women's Health Associates - Reston /ID# 217990, Reston, Virginia
  - Clinical Research Partners, LLC /ID# 216355, Richmond, Virginia
  - The Chronic Pelvic Pain Center of Northern VA /ID# 217630, Vienna, Virginia
  - Seattle Reproductive Medicine /ID# 213801, Seattle, Washington
  - West Virginia University /ID# 217664, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/elagolix_P16-836.pdf